CLINICAL TRIAL: NCT05400382
Title: Optimizing Mindfulness to Reduce Post-cesarean Pain and Prevent Postpartum Depression
Brief Title: Mindfulness to Reduce Post-cesarean Pain and Prevent Postpartum Depression
Acronym: MaMiDaPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of Pittsburgh Medical Center (Other); Southern Illinois University (Other); Arrowhead Regional Medical Center (Other); Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Principal Investigator, Sandraluz Lara-Cinisomo, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MaMiDaPP
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Depression, Unipolar; Pain, Postoperative
Keywords: postpartum; depression; pain; cesarean
MeSH Terms: conditions — Depressive Disorder; Pain, Postoperative; Depression; Pain | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Receiving mobile, self-guided mindfulness intervention
  Interventions: Behavioral: Mindfulness
- Treatment as usual with monitoring (No Intervention): Receiving treatment as usual with monitoring by study PI and investigators.

INTERVENTIONS:
Behavioral: Mindfulness — Meditation training to help reduce stress and reactivity to pain and other stressors.
  Other Names: Mindfulness meditation
  Arms: Mindfulness

SUMMARY:
This study will test the effect of a mobile mindfulness-based intervention on reducing post-cesarean delivery pain and preventing postpartum depression.

DETAILED DESCRIPTION:
This clinical trial will test the effect of a mobile mindfulness-based intervention on reducing post-cesarean delivery pain and preventing postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age, have a singleton pregnancy, score less than 10 on the Edinburgh Postnatal Depression Scale (EPDS; (Cox et al., 1987b), willing to participate in the eight-week intervention or be randomized to the TAUM condition, have no significant psychiatric disorders other than depression or anxiety (e.g., bipolar disorder, substance use disorder, etc.), have no chronic pain condition (e.g., fibromyalgia), and proficient in English or Spanish

Exclusion Criteria:

* Women who screen 10 or higher on the EPDS

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cis-gender women
Enrollment: 75 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Postpartum depression | 4 weeks - 6 months
  depressive symptoms EPDS 13 or higher

SECONDARY OUTCOMES:
Post-operative pain | 4 weeks - 6 months
  Post-cesarean delivery pain

IPD SHARING:
Plan to Share IPD: Undecided
To be determined